CLINICAL TRIAL: NCT05971238
Title: Characterization of Eye Movement Behaviour and Pupil Size Through Eye-tracking in Natural Outdoor and Indoor Scenes
Brief Title: Eye Movement Behaviour and Pupil Size in Natural Outdoor and Indoor Scenes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Collaborators: Max-Planck Institute for Biological Cybernetics (Other)
Responsible Party: Principal Investigator, Manuel Spitschan, Assistant Professor of Chronobiology & Health, Technical University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPI-TSCN-2023-NATURALEYE; 2023-231-S-KH (Other: Ethikkommission der Technischen Universität München)
Record Dates: First submitted 2023-06-05; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Light Sensitivity
MeSH Terms: conditions — Photophobia

STUDY DESIGN:
Intervention Model Description: All participants will be exposed to the same environmental conditions (same indoor and outdoor scenes for the same duration) and the captured eye-movement data of every participant will be of the same type. Participants will be exposed to different orders of scene sequences.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eye-tracking, pupillometry and scene rating indoors & outdoors (Experimental)
  Interventions: Other: Indoor vs. outdoor scenes

INTERVENTIONS:
Other: Indoor vs. outdoor scenes — Light conditions in indoor (artificial light) and outdoor (daylight) settings

SUMMARY:
In this study, the researchers will be using eye tracking and detailed lighting measurements to understand how different types of indoor and outdoor lighting affect the eye movements and pupil sizes of our participants. Participants will be paired up and undergo six eye tracking sessions, split across two appointments. Each appointment will involve viewing either indoor or outdoor scenes, and before each session, participants will spend time adapting to the lighting conditions. Overall, each participant will spend 24 minutes being tracked, and the entire study will take about 2-3 hours to complete. The investigators expect differences in eye movements and pupil size between indoor and outdoor scenes.

ELIGIBILITY:
Inclusion Criteria:

* No previous eye-surgeries or ocular impairments like anisometropia, amblyopia, strabism, cataract, watery eyes or hanging eye lids
* Normal or corrected-to-normal visual acuity (+3dpt. to -5dpt.)
* Normal colour vision
* Normal binocular vision

Exclusion Criteria:

* Any use of medications or drugs that influence photosensitivity or the ability to concentrate
* Excessive alcohol and/or drug use
* Presence of psychiatric disorders
* Poor sleep quality
* Diagnosed with epilepsy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Saccade frequency - Indoor scene 1 | Baseline
  Number per second [n/s]
Saccade frequency - Indoor scene 2 | Baseline
  Number per second [n/s]
Saccade frequency - Indoor scene 3 | Baseline
  Number per second [n/s]
Saccade frequency - Outdoor scene 1 | Baseline
  Number per second [n/s]
Saccade frequency - Outdoor scene 2 | Baseline
  Number per second [n/s]
Saccade frequency - Outdoor scene 3 | Baseline
  Number per second [n/s]
Saccade amplitude - Indoor scene 1 | Baseline
  Mean angular distance traveled [°]
Saccade amplitude - Indoor scene 2 | Baseline
  Mean angular distance traveled [°]
Saccade amplitude - Indoor scene 3 | Baseline
  Mean angular distance traveled [°]
Saccade amplitude - Outdoor scene 1 | Baseline
  Mean angular distance traveled [°]
Saccade amplitude - Outdoor scene 2 | Baseline
  Mean angular distance traveled [°]
Saccade amplitude - Outdoor scene 3 | Baseline
  Mean angular distance traveled [°]
Saccade velocity - Indoor scene 1 | Baseline
  Mean peak velocity [°/s]
Saccade velocity - Indoor scene 2 | Baseline
  Mean peak velocity [°/s]
Saccade velocity - Indoor scene 3 | Baseline
  Mean peak velocity [°/s]
Saccade velocity - Outdoor scene 1 | Baseline
  Mean peak velocity [°/s]
Saccade velocity - Outdoor scene 2 | Baseline
  Mean peak velocity [°/s]
Saccade velocity - Outdoor scene 3 | Baseline
  Mean peak velocity [°/s]
Fixation duration - Indoor scene 1 | Baseline
  Mean fixation duration [s]
Fixation duration - Indoor scene 2 | Baseline
  Mean fixation duration [s]
Fixation duration - Indoor scene 3 | Baseline
  Mean fixation duration [s]
Fixation duration - Outdoor scene 1 | Baseline
  Mean fixation duration [s]
Fixation duration - Outdoor scene 2 | Baseline
  Mean fixation duration [s]
Fixation duration - Outdoor scene 3 | Baseline
  Mean fixation duration [s]
Fixation frequency - Indoor scene 1 | Baseline
  Number per minute [n/min]
Fixation frequency - Indoor scene 2 | Baseline
  Number per minute [n/min]
Fixation frequency - Indoor scene 3 | Baseline
  Number per minute [n/min]
Fixation frequency - Outdoor scene 1 | Baseline
  Number per minute [n/min]
Fixation frequency - Outdoor scene 2 | Baseline
  Number per minute [n/min]
Fixation frequency - Outdoor scene 3 | Baseline
  Number per minute [n/min]
Pupil size - Indoor scene 1 | Baseline
  Mean pupil size [mm]
Pupil size - Indoor scene 2 | Baseline
  Mean pupil size [mm]
Pupil size - Indoor scene 3 | Baseline
  Mean pupil size [mm]
Pupil size - Outdoor scene 1 | Baseline
  Mean pupil size [mm]
Pupil size - Outdoor scene 2 | Baseline
  Mean pupil size [mm]
Pupil size - Outdoor scene 3 | Baseline
  Mean pupil size [mm]
Melanopic irradiance - Indoor scene 1 | Baseline
  Irradiance [W/(sqm*nm)]
Melanopic irradiance - Indoor scene 2 | Baseline
  Irradiance [W/(sqm*nm)]
Melanopic irradiance - Indoor scene 3 | Baseline
  Irradiance [W/(sqm*nm)]
Melanopic irradiance - Outdoor scene 1 | Baseline
  Irradiance [W/(sqm*nm)]
Melanopic irradiance - Outdoor scene 2 | Baseline
  Irradiance [W/(sqm*nm)]
Melanopic irradiance - Outdoor scene 3 | Baseline
  Irradiance [W/(sqm*nm)]
Photopic illuminance - Indoor scene 1 | Baseline
  Illuminance [lux]
Photopic illuminance - Indoor scene 2 | Baseline
  Illuminance [lux]
Photopic illuminance - Indoor scene 3 | Baseline
  Illuminance [lux]
Photopic illuminance - Outdoor scene 1 | Baseline
  Illuminance [lux]
Photopic illuminance - Outdoor scene 2 | Baseline
  Illuminance [lux]
Photopic illuminance - Outdoor scene 3 | Baseline
  Illuminance [lux]

SECONDARY OUTCOMES:
Subjective scene ratings - Indoor scene 1 | Baseline
  * Unabbreviated scale titles (1)., min. and max, values (2.), score assessment (3.):
  * 1. "How beautiful is this scene to you?" 2. "1 = not beautiful at all; 10 = extremely beautiful" 3. No better or worse outcome
  * 1. "How would you rate the brightness of this scene?" 2. "1 = dimly lit room; 10 = bright sunny day" 3. No better or worse outcome
  * 1. "How visually comfortable did you find this scene?" 2. "1 = No discomfort; 10 = Very uncomfortable" 3. No better or worse outcome
  * 1. "How would you rate the complexity of the scene (e.g. colour contrasts, different object identities, moving objects)?" 2. "1 = very simple; 10 = Very complex" 3. No better or worse outcome
  * 1. "How sleepy do you currently feel" 2. "1 = Extremely alert; 10 = Extremely sleep, can't keep awake" 3. Lower score is better
Subjective scene ratings - Indoor scene 2 | Baseline
  * Unabbreviated scale titles (1)., min. and max, values (2.), score assessment (3.):
  * 1. "How beautiful is this scene to you?" 2. "1 = not beautiful at all; 10 = extremely beautiful" 3. No better or worse outcome
  * 1. "How would you rate the brightness of this scene?" 2. "1 = dimly lit room; 10 = bright sunny day" 3. No better or worse outcome
  * 1. "How visually comfortable did you find this scene?" 2. "1 = No discomfort; 10 = Very uncomfortable" 3. No better or worse outcome
  * 1. "How would you rate the complexity of the scene (e.g. colour contrasts, different object identities, moving objects)?" 2. "1 = very simple; 10 = Very complex" 3. No better or worse outcome
  * 1. "How sleepy do you currently feel" 2. "1 = Extremely alert; 10 = Extremely sleep, can't keep awake" 3. Lower score is better
Subjective scene ratings - Indoor scene 3 | Baseline
  * Unabbreviated scale titles (1)., min. and max, values (2.), score assessment (3.):
  * 1. "How beautiful is this scene to you?" 2. "1 = not beautiful at all; 10 = extremely beautiful" 3. No better or worse outcome
  * 1. "How would you rate the brightness of this scene?" 2. "1 = dimly lit room; 10 = bright sunny day" 3. No better or worse outcome
  * 1. "How visually comfortable did you find this scene?" 2. "1 = No discomfort; 10 = Very uncomfortable" 3. No better or worse outcome
  * 1. "How would you rate the complexity of the scene (e.g. colour contrasts, different object identities, moving objects)?" 2. "1 = very simple; 10 = Very complex" 3. No better or worse outcome
  * 1. "How sleepy do you currently feel" 2. "1 = Extremely alert; 10 = Extremely sleep, can't keep awake" 3. Lower score is better
Subjective scene ratings - Outdoor scene 1 | Baseline
  * Unabbreviated scale titles (1)., min. and max, values (2.), score assessment (3.):
  * 1. "How beautiful is this scene to you?" 2. "1 = not beautiful at all; 10 = extremely beautiful" 3. No better or worse outcome
  * 1. "How would you rate the brightness of this scene?" 2. "1 = dimly lit room; 10 = bright sunny day" 3. No better or worse outcome
  * 1. "How visually comfortable did you find this scene?" 2. "1 = No discomfort; 10 = Very uncomfortable" 3. No better or worse outcome
  * 1. "How would you rate the complexity of the scene (e.g. colour contrasts, different object identities, moving objects)?" 2. "1 = very simple; 10 = Very complex" 3. No better or worse outcome
  * 1. "How sleepy do you currently feel" 2. "1 = Extremely alert; 10 = Extremely sleep, can't keep awake" 3. Lower score is better
Subjective scene ratings - Outdoor scene 2 | Baseline
  * Unabbreviated scale titles (1)., min. and max, values (2.), score assessment (3.):
  * 1. "How beautiful is this scene to you?" 2. "1 = not beautiful at all; 10 = extremely beautiful" 3. No better or worse outcome
  * 1. "How would you rate the brightness of this scene?" 2. "1 = dimly lit room; 10 = bright sunny day" 3. No better or worse outcome
  * 1. "How visually comfortable did you find this scene?" 2. "1 = No discomfort; 10 = Very uncomfortable" 3. No better or worse outcome
  * 1. "How would you rate the complexity of the scene (e.g. colour contrasts, different object identities, moving objects)?" 2. "1 = very simple; 10 = Very complex" 3. No better or worse outcome
  * 1. "How sleepy do you currently feel" 2. "1 = Extremely alert; 10 = Extremely sleep, can't keep awake" 3. Lower score is better
Subjective scene ratings - Outdoor scene 3 | Baseline
  * Unabbreviated scale titles (1)., min. and max, values (2.), score assessment (3.):
  * 1. "How beautiful is this scene to you?" 2. "1 = not beautiful at all; 10 = extremely beautiful" 3. No better or worse outcome
  * 1. "How would you rate the brightness of this scene?" 2. "1 = dimly lit room; 10 = bright sunny day" 3. No better or worse outcome
  * 1. "How visually comfortable did you find this scene?" 2. "1 = No discomfort; 10 = Very uncomfortable" 3. No better or worse outcome
  * 1. "How would you rate the complexity of the scene (e.g. colour contrasts, different object identities, moving objects)?" 2. "1 = very simple; 10 = Very complex" 3. No better or worse outcome
  * 1. "How sleepy do you currently feel" 2. "1 = Extremely alert; 10 = Extremely sleep, can't keep awake" 3. Lower score is better
Geographical scene location - Indoor scene 1 | Baseline
  Longitude and latitude [°]
Geographical scene location - Indoor scene 2 | Baseline
  Longitude and latitude [°]
Geographical scene location - Indoor scene 3 | Baseline
  Longitude and latitude [°]
Geographical scene location - Outdoor scene 1 | Baseline
  Longitude and latitude [°]
Geographical scene location - Outdoor scene 2 | Baseline
  Longitude and latitude [°]
Geographical scene location - Outdoor scene 3 | Baseline
  Longitude and latitude [°]
Ambient temperature - Indoor scene 1 | Baseline
  Temperature [°C]
Ambient temperature - Indoor scene 2 | Baseline
  Temperature [°C]
Ambient temperature - Indoor scene 3 | Baseline
  Temperature [°C]
Ambient temperature - Outdoor scene 1 | Baseline
  Temperature [°C]
Ambient temperature - Outdoor scene 2 | Baseline
  Temperature [°C]
Ambient temperature - Outdoor scene 3 | Baseline
  Temperature [°C]

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Spitschan, PhD, Principal Investigator — Technical University of Munich & Max Planck Institute for Biological Cybernetics
Locations (1):
- Max Planck Institute for Biological Cybernetics, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Yes